CLINICAL TRIAL: NCT06670157
Title: Detachable Clip-assisted Endoscopic Cyanoacrylate Injection in the Treatment of Gastric Varices Under X-ray Perspective
Brief Title: Detachable Clip-assisted Endoscopic Cyanoacrylate Injection in the Treatment of Gastric Varices
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yu Chang (Other)
Responsible Party: Sponsor-Investigator, Yu Chang, student, Nanjing University of Traditional Chinese Medicine
Organization: Nanjing University of Traditional Chinese Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DZQH-KYLL-24-16
Record Dates: First submitted 2024-10-31; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Gastric Varices Bleeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Detachable Clip-assisted (Experimental): After the varicose vessel is closed with a removable titanium clamp, the more varicose target vessel is located，After the varicose vessels basically disappeared under the endoscope, the removable titanium clamp was removed
  Interventions: Other: Detachable Clip

INTERVENTIONS:
Other: Detachable Clip — After the varicose vessels basically disappeared under the endoscope, the removable titanium clamp was removed

SUMMARY:
A single-arm exploratory clinical study design was used to evaluate the safety and efficacy of a "modified sandwich injection" of tissue glue assisted by a detachable clip for the treatment of gastric varicose veins.

ELIGIBILITY:
Inclusion Criteria:

* The subject voluntarily signs the informed consent for this experiment; According to clinical manifestation, laboratory examination, imaging examination, or liver biopsy in the diagnosis of liver cirrhosis patients; The endoscopy diagnosed gastric varices (gastroesophageal varices, gastroesophageal varices type 2 or type 1 isolated gastric varices type 1); High risk of gastric varices or has a history of gastric varices bleeding. The initial fluid resuscitation patients before or after the recovery hemodynamic stability; The age of 18 years old or more.

Exclusion Criteria:

* < 18 years old; Regional portal hypertension; Always have a liver transplant, via the jugular intrahepatic portal vein system bypass or splenectomy combined varices cut-out art history; A concurrent hepatorenal syndrome and/or multiple organ failure; Significant impact on survival of malignant tumor; Pregnancy or lactation; A known allergy to iodine.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Rebleeding rate at 6 weeks after treatment for gastric fundus varicose veins in cirrhosis | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: ji xuan, doctor, Principal Investigator — Eastern Theater General Hospital
Locations (1):
- Eastern Theater General Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR